CLINICAL TRIAL: NCT03740022
Title: Assessment of the Results of Combined Anterolateral Ligament (ALL) + Antero Crusader Ligament (ACL) Plasty Compared to Classical KJ Plasty in Isolated ACL Ruptures
Brief Title: ACL Versus ALL + ACL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascopharm Groupe Novasco (Other)
Collaborators: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-A00144-47
Record Dates: First submitted 2016-11-29; First posted 2018-11-14 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Anterior Cruciate Ligament Injury; Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACL plasty (Active Comparator): The surgical procedure consists of a ligamentoplasty of the antero crusader ligament (ACL) with the patellar tendon according to a conventional arthroscopic procedure.
  Interventions: Procedure: ACL plasty
- ACL + ALL plasty (Experimental): The surgical procedure consists of a hamstring ligamentoplasty (DIDT) of the antero crusader ligament (ACL) and anterolateral ligament (ALL) according to a published arthroscopic procedure.
  Interventions: Procedure: ACL + ALL plasty

INTERVENTIONS:
Procedure: ACL plasty — standard ligamentoplasty by Kenneth Jones
  Arms: ACL plasty
Procedure: ACL + ALL plasty — standard ligamentoplasty and anterolateral plasty
  Arms: ACL + ALL plasty

SUMMARY:
The aim of the study is to show a reduction of a re-rupture rate with an ACL (antero crusader ligament) + ALL (anterolateral ligament) combined technique compared to a classical Kenneth-Jones ACL (antero crusader ligament) reconstruction technique.

DETAILED DESCRIPTION:
The aim is to evaluate the rate of re-rupture and to analyze knee function through scores analysis as International Knee Documentation Committee Subjective Knee (IKDC), Knee injury and osteoarthritis outcome score (KOOS), Lysholm-Tegner, and by objective measurements of laximetry and rotation.

This study should include 2 groups of 296 patients with isolated ACL (antero crusader ligament) with clinical rotation :

* operated by a conventional patellar tendon technique (first group)
* operated by a technique combining a ALL (anterolateral ligament) and ACL plasty for the second group

ELIGIBILITY:
Inclusion Criteria:

* Patients with total isolated antero crusader ligament (ACL) rupture who are candidates for surgical reconstruction
* Patients between 18 and 35 years old
* Patients with weekly sporting activities
* Patients with chronic rotatory instability with a positive pivot shift
* Patients who have been informed and do not object the research

Exclusion Criteria:

* Patients with multi-ligament knee involvement
* Patients under 18 years old or over 35 years old
* Patients with a BMI of under 18.5 or over 30
* Patients with any contraindication to general anaesthesia
* Professional sportsmen/women
* Patients with congenital malformation or a rheumatic disease
* Patients with repeated antero crusader ligament (ACL) rupture
* Patients with serious ligament disease in the contralateral knee
* Patients who refuse to take part in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 592 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Ligament re-rupture rate | 3 years
  Clinical instability, laximetry, IRM

SECONDARY OUTCOMES:
International Knee Documentation Committee Subjective Knee (IKDC) clinical score | preoperatively, 1 year and 3 years
  International Knee Documentation Committee Subjective Knee allows a subjective assessment including symptoms, activity and knee function; is scored by summing the scores for the individual items and then transforming the score to a scale that ranges from 0 to 100 (no limitation with activities of daily living or sports activities and the absence of symptoms)
Tegner Lysholm score | Preoperatively, 1 year and 3 years
  Specific knee questionnaire : patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Rolimeter test | pre-operatively, 6 months, 1 year and 3 years
  Antero-posterior laximetry
KiRA test | preoperatively, 6 months and 3 years
  Rotatory laximetry
Knee radiography | preoperatively and 3 years
  Development of osteoarthritis signs
Knee injury and osteoarthritis outcome score (KOOS) clinical score | preoperative, 1 year and 3 years
  Knee injury and osteoarthritis outcome score is a specific knee questionnaire which evaluates : pain, symptoms, knee function in daily life, knee function in sport practice and quality of life. Scale : None (0) Mild Moderate Severe Extreme (4) Each subscale score is calculated independently. Calculate the mean score of the individual items of each subscale and divide by 4. Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz - Centre Paul Santy, Lyon, France

REFERENCES:
- [Derived] Sonnery-Cottet B, Carrozzo A, Poilvache H, Fayard JM, Freychet B, Thaunat M, Vieira TD, Saithna A; Santy Orthopedic Center Group. Anterior cruciate ligament reconstruction combined with anterolateral ligament reconstruction using hamstring autograft versus anterior cruciate ligament reconstruction using bone-patellar tendon-bone autograft: a randomised controlled trial with 5-year follow-up. Lancet Reg Health Eur. 2025 Dec 20;62:101561. doi: 10.1016/j.lanepe.2025.101561. eCollection 2026 Mar. PMID 41536854
- [Derived] Sonnery-Cottet B, Pioger C, Vieira TD, Franck F, Kajetanek C, Fayard JM, Thaunat M, Saithna A. Combined ACL and Anterolateral Reconstruction Is Not Associated With a Higher Risk of Adverse Outcomes: Preliminary Results From the SANTI Randomized Controlled Trial. Orthop J Sports Med. 2020 May 1;8(5):2325967120918490. doi: 10.1177/2325967120918490. eCollection 2020 May. PMID 32490026